CLINICAL TRIAL: NCT05054231
Title: Immunological Profile for Patients Treated With CAR-T Cells
Acronym: SI-CART
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Paoli-Calmettes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SI-CART-IPC 2019-006
Record Dates: First submitted 2020-07-28; First posted 2021-09-23 (Actual); Last update posted 2021-10-15 (Actual); Status verified 2021-10

CONDITIONS: Hematologic Neoplasms
Keywords: CAR-T cells; Immunological Profile
MeSH Terms: conditions — Hematologic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient treated with CAR-T cells (Experimental)
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood samples collection: at Day (D)-6 and D0 before CAR-T cells injection, post injection at Day (D)3, D5,D7, D9, D11, D14, D18, D 21, Month 2 and Month 12 post injection.

SUMMARY:
In the frame of Si-CART study, blood will be collected from patients treated with CAR-T cells: before (at Day (D)-6 and D0 before cells injection), post infusion at D3, D5,D7, D9, D11, D14, D18, D 21, Month (M) 2 and M12 post injection.

A cerebrospinal fluid sample will also be collected if a Cerebrospinal Fluid Analysis Lumbar puncture is performed

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Planned injection of CAR-T cells within the scope of marketing authorization
* Signed informed consent
* French social security affiliation

Exclusion Criteria:

* Pregnant women, or women of childbearing potential (without medically acceptable contraception) or breastfeeding women.
* Patient in emergency situation, adult under legal protection (patient placed under tutorship, curatorship, or judicial protection) or unable to give his consent
* Impossibility to comply with trial medical follow-up for geographic, social or psychological reasons

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2021-10-05 (Estimated); Primary Completion 2025-10-05 (Estimated); Study Completion 2026-10-05 (Estimated)

PRIMARY OUTCOMES:
Correlation between serum markers and adverse events at 1 year of the CAR-T cells infusion | 1 year after T cells infusion
  Serum concentration of cytokines in relation to adverse events

SECONDARY OUTCOMES:
CAR-T cells rate from infusion to one year after CAR-T cells infusion | From CAR-T cells infusion to one year
  Flow cytometry
Number of participants with a relapse | From CAR-T cells infusion to one year
  Relapse rate from CAR-T cells infusion to one year
Number of participants with a cytokine release syndrome | From CAR-T cells infusion to one year
  Cytokine release syndrome from CAR-T cells infusion to one year

CONTACTS AND LOCATIONS:
Locations (1):
- Institut Paoli-Calmettes, Marseille, France

IPD SHARING:
Plan to Share IPD: No